CLINICAL TRIAL: NCT03798132
Title: Imaging Evaluation of Peritoneal Carcinomatosis Extent
Brief Title: Peritoneal Carcinomatosis Extent Evaluation: Radiologic, Laparoscopic and Pathologic.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shimaa Abdalla Ahmed (Other)
Responsible Party: Sponsor-Investigator, Shimaa Abdalla Ahmed, lecturer of radiodiagnosis, South Egypt Cancer Institute
Organization: South Egypt Cancer Institute (Other)
Other Study IDs: SouthECI
Record Dates: First submitted 2019-01-07; First posted 2019-01-09 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Peritoneal Carcinomatosis
Keywords: Ovarian Neoplasms, Laparoscopy, Cytoreduction Surgical Procedures.
MeSH Terms: conditions — Peritoneal Neoplasms; Ovarian Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: laparoscopy — evaluation of peritoneal carcinomatosis by laparoscopy

SUMMARY:
pathologically proved ovarian cancer patients that underwent contrast enhanced abdomino-pelvic CT and diagnostic laparoscopy before cytoreductive surgery (CRS) will be included in the study. Calculation of PCI (peritoneal cancer index) using Sugarbaker's method, peritoneal carcinomatosis extent will be categorized into low, moderate and large. Agreement in general and in each category between CT, laparoscopy, surgery and pathology will be assessed using kappa agreement.

DETAILED DESCRIPTION:
we will search medical records of primary ovarian cancer patients underwent CT abdomen, laparoscopy followed by cytoreductive surgery to calculate peritoneal carcinomatosis extent by each modality.

Regional PCI was calculated in each of the 13 anatomical abdominopelvic regions, then total PCI by summation of the lesion size score, it ranged from 0 to 39. Categorization of peritoneal carcinomatosis was classified into 3 categories low if PCI < 10, moderate if 10-20, and large if >20.

ELIGIBILITY:
Inclusion Criteria:pathologically proved ovarian cancer patients underwent contrast enhanced abdominopelvic CT and diagnostic laparoscopy before cytoreductive surgery -

Exclusion Criteria:recurrent ovarian cancer

-

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pathologically proved ovarian cancer patients recived cytoreductive surgery and underwent preoperative CT and diagnostic laparoscopy
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-06-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
peritoneal carcinomatosis | one year
  Agreement in general and in each category between CT, laparoscopy, surgery and pathology was assessed using kappa agreement.

SECONDARY OUTCOMES:
surgical decision making. | one year
  correlation of peritoneal carcinomatosis categorization with surgical decision

CONTACTS AND LOCATIONS:
Locations (1):
- South Egypt Cancer Institute, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fagotti A, Ferrandina G, Fanfani F, Garganese G, Vizzielli G, Carone V, Salerno MG, Scambia G. Prospective validation of a laparoscopic predictive model for optimal cytoreduction in advanced ovarian carcinoma. Am J Obstet Gynecol. 2008 Dec;199(6):642.e1-6. doi: 10.1016/j.ajog.2008.06.052. Epub 2008 Sep 17. PMID 18801470